CLINICAL TRIAL: NCT06102759
Title: Phase II Clinical Study of Adebrelimab and Fruquintinib Combined With Paclitaxel/Albumin Paclitaxel for Second-line Treatment of Advanced Gastric Cancer After First-line Treatment With PD-1 Antibody Failed
Brief Title: Adebrelimab and Fruquintinib Combined With Paclitaxel/Albumin Paclitaxel for Advanced Gastric Cancer After PD-1 Antibody Failed
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJMUCH-GI-GC04
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; second-line treatment; Adebrelimab; Fruquintinib; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adebrelimab, Fruquintinib combined with paclitaxel: Fruquintinib 4mg d1-14, q3w Paclitaxel 150mg/m2, d1, q3w / Albumin paclitaxel 125mg/m2, d1, d8, q3w PD-L1 antibody (Adebrelimab) 20 mg/kg, d1, q3w
  Interventions: Drug: Adebrelimab，Fruquintinib

INTERVENTIONS:
Drug: Adebrelimab，Fruquintinib — Adebrelimab，Fruquintinib combined with chemotherapy

SUMMARY:
This is a prospective, single-center, open, single-arm clinical study to observe and evaluate the efficacy and safety of Fruquintinib and Adebrelimab combined with paclitaxel/albumin paclitaxel for second-line treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
Since the first-line ICIs application of gastric cancer is mainly PD-1 antibody, this study intends to screen first-line patients exposed to PD-1 antibody and with long survival (PFS longer than 9 months) to receive second-line PD-L1 antibody for re-challenge and combine with Fruquintinib and paclitaxel to explore whether it can further increase the effect of second-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. The ECOG score is 0-1 and does not deteriorate within 7 days.
3. Patients with histologically confirmed, metastatic, or unresectable locally advanced gastric cancer or GEJ adenocarcinoma.
4. Previously received one systemic chemotherapy regimen for this cancer and progressed; Or have received adjuvant chemotherapy, but have disease progression or recurrence within 6 months after the end of treatment.
5. First-line exposure to PD-1 antibodies and first-line treatment of PFS greater than 9 months.
6. Measurable lesions that meet RECIST 1.1 criteria.
7. Have adequate organ and bone marrow function, laboratory tests meet the following requirements:

   1. HGB≥90g/L;
   2. NEUT≥1.5×10^9/L;
   3. PLT ≥80×10^9/L;
   4. TBIL≤1.5 times upper limit of normal value (ULN);
   5. ALT and AST≤2.5 x ULN; In liver metastasis, ALT and AST≤5×ULN;
   6. Endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
   7. Urinary protein < (++), or 24-hour urinary protein volume < 1.0 g.
8. Normal coagulation function, no active bleeding

   1. International standardized ratio INR≤1.5;
   2. Partial thromboplastin time APTT≤1.5 ULN.
9. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days prior to enrollment and voluntarily use an appropriate method of contraception during the observation period and within 8 weeks after the last dose of the study drug; For men, they should be surgically sterilized or consent to an appropriate method of contraception during the observation period and for 8 weeks after the last administration of the study drug.
10. Expected survival ≥3 months.
11. Patients voluntarily joined the study and signed an informed consent form (ICF).
12. It is expected that the compliance is good, and the efficacy and adverse reactions can be followed up according to the protocol requirements.

Exclusion Criteria:

1. Previous treatment with VEGFR inhibitors;
2. Previously received paclitaxel therapy (except for those who received paclitaxel therapy in neoadjuvant or adjuvant therapy, and the treatment ended more than 6 months after the disease progression);
3. Receive live vaccine within 4 weeks prior to enrollment or possibly during the study period;
4. Had active autoimmune disease or history of autoimmune disease within 4 weeks prior to enrollment;
5. Previously received allogeneic bone marrow transplantation or organ transplantation;
6. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg;
7. Had any disease or condition affecting drug absorption before enrollment, or the patient could not take drugs orally;
8. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unexcised tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
9. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis, or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months;
10. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure > Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;
11. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);
12. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or > 2000 IU/ mL); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL);
13. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
14. The patients considered by the investigators to be unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer that failed first-line treatment with PD1 antibody
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Time from the start of treatment to the progression of the disease

SECONDARY OUTCOMES:
Disease Control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR,PR and SD
The Overall Response Rate | Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The proportion of CR and PR
Overall survival | From date of randomization until the date of death from any cause or the last visit date, whichever came first, assessed up to 60 months
  Time from the start of treatment to the occurrence of death

CONTACTS AND LOCATIONS:
Overall Officials: Ting Deng, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Sharma P, Hu-Lieskovan S, Wargo JA, et al. Primary, Adaptive, and Acquired Resistance toCancer Immunotherapy. Cell 2017; 168: 707-723. 2. Teng MW, Ngiow SF, Ribas A, et al. Classifying Cancers Based on T-cell Infiltration and PD-L1.Cancer Res 2015; 75: 2139-45. 3. Olson DJ, Eroglu Z, Brockstein B, et al. Pembrolizumab Plus Ipilimumab Following Anti-PD1/L1 Failure in Melanoma. J Clin Oncol 2021; 39: 2647-2655. 4. Pires da Silva I, Ahmed T, Reijers ILM, et al. Ipilimumab alone or ipilimumab plus anti-PD-1therapy in patients with metastatic melanoma resistant to anti-PD-(L)1 monotherapy: a multicentre,retrospective, cohort study. Lancet Oncol 2021; 22: 836-847. 5. Zaremba A, Eggermont AMM, Robert C, et al. The concepts of rechallenge and retreatmentwith immune checkpoint blockade in melanoma patients. Eur J Cancer 2021; 155: 268-280. 6. Yang K, Li J, Sun Z, et al. Retreatment with immune checkpoint inhibitors in solid tumors: asystematic review. Ther Adv Med Oncol 2020; 12: 1758835920975353. 7. Vera Aguilera J, Paludo J, McWilliams RR, et al. Chemo-immunotherapy combination afterPD-1 inhibitor failure improves clinical outcomes in metastatic melanoma patients. Melanoma Res2020; 30: 364-375. 8. Giaj Levra M, Cotte FE, Corre R, et al. Immunotherapy rechallenge after nivolumabtreatment in advanced non-small cell lung cancer in the real-world setting: A national data baseanalysis. Lung Cancer 2020; 140: 99-106. 9. Kitagawa S, Hakozaki T, Kitadai R, et al. Switching administration of anti-PD-1 and anti-PD-L1antibodies as immune checkpoint inhibitor rechallenge in individuals with advanced non-small celllung cancer: Case series and literature review. Thorac Cancer 2020; 11: 1927-1933. 10. Takahara Y, Tanaka T, Ishige Y, et al. Efficacy and predictors of rechallenge with immunecheckpoint inhibitors in non-small cell lung cancer. Thorac Cancer 2022; 13: 624-630. 11. Zhang Y, Wang ZX, Shen L, et al. A phase Ib/II study of fruquintinib in combination withpaclitaxel as the second-line therapy for advanced gastric cancer. Cancer Commun (Lond) 2023; 43:150-153.